CLINICAL TRIAL: NCT05477680
Title: Intraoperative Brain Shift Calculation Study: a Prospective, Single Arm Clinical Trial
Brief Title: Intraoperative Brain Shift Calculation Study
Acronym: BRASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Alexander Dmitriev, Principal Investigator, Sklifosovsky Institute of Emergency Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9e
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tumor, Brain; Cavernoma; Arteriovenous Malformations; Intracerebral Hematoma
Keywords: brain shift; tumor; cavernoma; arteriovenous malformation; intracerebral hematoma
MeSH Terms: conditions — Brain Neoplasms; Hemangioma, Capillary; Arteriovenous Malformations; Cerebral Hemorrhage; Neoplasms | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery (Experimental): Removing different brain lesions using neuronavigation
  Interventions: Device: Navigation-guided surgery

INTERVENTIONS:
Device: Navigation-guided surgery — Surgeon removes brain lesions and assesses brain shift with neuronavigation

SUMMARY:
The purpose of the study is to calculate magnitude, type of intraoperative brain shift and assess possibility of it's prediction.

DETAILED DESCRIPTION:
Brain shift is the main natural cause of major navigation imprecision. Despite numerous attempts no trials showed a possibility to calculate and predict it's value although some patterns were found. Some modern navigational features allow to partially resolve this problem. Manual shift correction allows to displace brain structures but can only be used if brain shift is linear. Intraoperative computed tomography (CT) and magnetic resonance imaging (MRI) allow to update navigational data but violate surgical workflow and cannot display brain tissue in real time. Intraoperative sonography has poorer quality, limited observe volume and lengthy learning curve.

The purpose of the study is to calculate magnitude, type of intraoperative brain shift and assess possibility of it's prediction.

For each patient a surgeon intraoperatively will assess location of brain surface, various intracranial structures and lesion margins during surgery. Postoperatively these data will be compared to lesion's characteristics, patient's state and intraoperative features.

ELIGIBILITY:
Inclusion Criteria:

* all intracranial tumors
* cavernomas
* arteriovenous malformations
* spontaneous (non-traumatic) intracerebral hemorrhages
* traumatic intracerebral hemorrhages
* supratentorial localization
* newly diagnosed
* age 18-100 years
* stable hemodynamics
* error of patient registration in neuronavigation no more than 2 mm

Exclusion Criteria:

* rapid cerebral dislocation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Brain shift (in millimeters) | Intraoperatively
  Maximal difference between disposition of different brain structures in preoperative scans and it's real intraoperative location

SECONDARY OUTCOMES:
Karnofsky Performance status in percents | within 10 days after surgery
  Assesses patients' possibilities to self-service
Cerebral complications | From admission to intensive care unit after surgery till hospital discharge, up to 365 days
  Which cerebral complications arose after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dmitriev, MD, Principal Investigator — Sklifosovsky Institute of Emergency Care
Locations (1):
- Sklifosovsky Institute of Emergency Care, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No